CLINICAL TRIAL: NCT05620797
Title: Immediate Versus Delayed Loading for Immediately Inserted Implants Retaining Mandibular Complete Overdenture
Brief Title: Immediate Versus Delayed Loading for Implants Retaining Mandibular Complete Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: implant_86_2018
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Bone Loss; Dental Implant
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate loading implants (Experimental)
  Interventions: Other: Immediate loading of the implants
- Delayed loading implants (Active Comparator)
  Interventions: Other: Delayed loading of the implant

INTERVENTIONS:
Other: Immediate loading of the implants — Patients of this group will be rehabilitated by implant-retained mandibular overdenture with immediate loading of the implants as opposed to conventional maxillary complete dentures.
  Arms: Immediate loading implants
Other: Delayed loading of the implant — Patients of this group will be rehabilitated by implant retained mandibular overdenture with delayed loading of the implants (after 3 months) opposed by conventional maxillary complete dentures
  Arms: Delayed loading implants

SUMMARY:
The aim of this study will be to compare the amount of marginal bone height changes between immediate and delayed loading for immediately inserted implants used as abutments of mandibular overdenture.

ELIGIBILITY:
Inclusion Criteria:

* Patient having two standing mandibular canines with compromised prognosis (which indicted for extraction, without any preapical lesions nor acute infection) and have an adequate labial bone thickness.
* Patient having opposing completely edenteolous maxilla.
* Patients having normal maxilla-mandibular relationship and sufficient inter arch distance was insured by through tentative jaw relation record.
* Patients with good oral hygiene.
* Enough bone volume for implants in the interforaminal region (adequate bone quality and quantity)

Exclusion Criteria:

* Mental disorder patients who are not capable of making a decision or narcotic drug addicts.
* Patients with Tempro-Mandibular Joint disorders
* Patients undergoing radiotherapy or chemotherapy
* Patients with systemic diseases affecting bone metabolism
* Uncooperative patients who have no understanding of the need of a regular follow-up.
* Patient with pathological defects in the areas of implant insertion.
* Vulnerable group as prisoners, mentally retarded patients.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males only
Enrollment: 14 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in bone loss | at 3 months, 6 months, 9 months, 12 months
  Every 3 months all patients were recalled for assessment of marginal bone loss. The assessment was done using digital periapical radiograph Ezsensor (Vatech intraoral radiographic sensor, Vatech, South Korea) and the technique of radiograph was paralleling technique using sensor holder (TROLLBYTE PLUS, TROLLDENTAL, UK) to ensure same position of cone through subsequent follow-up exposures

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Faculty of Dentistry, Cairo, Egypt